CLINICAL TRIAL: NCT03977350
Title: A Blind, Observational, Prospective, Multi -Center, One Arm, Study on the Association Between qEEG Measure and Post-Operative Cognitive Dysfunction (POCD) and Postoperative Delirium (POD)
Brief Title: Association Between qEEG Measure and Post-Operative Cognitive Dysfunction (POCD) and Postoperative Delirium (POD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuroindex Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLD5
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients over 65 years undergoing heart surgery: Patients over 65 years undergoing heart surgery under anesthesia, EEG monitored
  Interventions: Device: EEG monitoring

INTERVENTIONS:
Device: EEG monitoring — EEG monitoring under general anesthesia

SUMMARY:
Cognitive complications after major surgery are a common phenomenon. The incidence of Postoperative Cognitive Dysfunction (POCD), may vary from 5% to 25% in adult patients, depending on different risk factors. Age has been strongly associated with cognitive complications. POCD is a prolonged decline in cognitive function that appears after surgery as compared with preoperative functions. In order to classify evaluate POCD, it requires at least 2 measurements. A baseline, completed before surgery and a second measurement, post surgery.

In light of the high prevalence of POCD and the difficulties in its prediction, NeuroIndex has developed a quantitative EEG system and software that aim to produces risk predictor index (IS) for POCD. This study aims to evaluate the relationship between the software produced predictor index and the actual POCD events. The qEEG will be monitored during the surgery in addition to the routine clinical practice in operating rooms.

POCD will be evaluated using Montreal Cognitive Assessment test (MoCA) prior and post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 65 or above.
* Subjects with American Society of Anesthesiologists physical status I-III.
* Subjects who are intended to undergo cardiac surgery (CABG or valve replacement) under general anesthesia.
* Surgical procedures scheduled for over 30 minutes.
* Lack of significant hearing disturbances.
* Subjects with ability to read and understand the consent form.

Exclusion Criteria:

* Significant visual impairment so that the pictures of the confusion assessment method could not be interpreted to accurately test to assess delirium.
* Profound dementia or aphasia that interfered with the assessment of cognitive dysfunction (positive delirium in CAM-ICU).
* Patients with a history of stroke.
* Any documented major neurologic or psychiatric dysfunction.
* Pregnant women.
* Long term use of sedative-hypnotic drugs and antidepressant drug.
* Subjects with scalp or skull abnormalities (s/p brain surgery, cranial implants).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will consist of male and female adults undergoing cardiac surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The qEEG parameter IS correlation with POCD | 1 week following surgery
  The qEEG parameter IS, which range between 0 and 1, where higher scores are more favorable than lower scores will be evaluated for its correlation with POCD that will be measured by Montreal Cognitive Assessment (MoCA)

CONTACTS AND LOCATIONS:
Overall Officials: Dror Leviner, Dr., Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No